CLINICAL TRIAL: NCT02316834
Title: POSITION: A Pilot Study of Induction PARP Inhibition in Ovarian Cancer
Brief Title: Talazoparib in Determining Genetic Effects on Disease Response in Patients With Advanced Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Acronym: POSITION
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0474; NCI-2014-02608 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0474 (Other: M D Anderson Cancer Center); P30CA016672 (NIH); P50CA083639 (NIH)
Record Dates: First submitted 2014-12-05; First posted 2014-12-15 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Fallopian Tube Serous Adenocarcinoma; High Grade Ovarian Serous Adenocarcinoma; Ovarian Mass; Primary Peritoneal Serous Adenocarcinoma; Stage III Fallopian Tube Cancer AJCC v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

ARMS (1):
- BMN 673 (Experimental)
  Interventions: Other: Laboratory Biomarker Analysis; Drug: BMN 673

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: BMN 673 — BMN673 given at a dose of 1 mg orally once daily.
  Participants begin taking BMN 673 tablets by mouth every day, starting on the day of scheduled laparoscopy. Participants take the study drug for at least 7 days before scheduled tumor reduction surgery.
  Other Names: TALAZOPARIB

SUMMARY:
This pilot early phase I trial studies talazoparib to determine if certain characteristics of the deoxyribonucleic acid (DNA) affect how the disease responds to therapy in patients with ovarian, fallopian tube, or primary peritoneal cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Studying samples of tissue in the laboratory from patients receiving talazoparib may help doctors learn more about the effects of talazoparib on cells and may help doctors understand how well patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore basal levels and effects of talazoparib (BMN 673) on DNA copy number, loss of heterozygosity and mutation, and level of ribonucleic acid (RNA) and protein expression (together described as "molecular results") in homologous recombination-related pathways before and after treatment in women with primary advanced high grade serous ovarian, fallopian tube, or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. To correlate molecular results to clinical endpoints including response and survival.

II. To correlate molecular results to pathologic endpoints including tumor volume and apoptosis.

III. To compare DNA copy number and level of RNA and protein expression in homologous recombination-related pathways in tissue from patients treated with BMN 673 to those untreated with BMN 673 in the preoperative period.

IV. To determine the toxicity of daily BMN 673 given preoperatively, with a focus on postoperative wound healing.

V. To determine feasibility of daily BMN 673 given preoperatively.

OUTLINE:

Patients receive talazoparib orally (PO) once daily (QD) for up to 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with presumed advanced-stage high grade serous ovarian, fallopian tube, or primary peritoneal carcinoma, based on the presence of carcinomatosis, and/or elevated cancer antigen 125 (CA125), and/or ovarian mass(es), or at the discretion of the treating physician
* Medically able to undergo primary cytoreductive surgery, at least 7 days and up to 28 days after starting study drug, as determined by treating physician
* No prior therapy for high-grade serous ovarian, fallopian tube, or primary peritoneal carcinoma
* Patients must be able to swallow and tolerate oral medications and not have gastrointestinal illnesses that would preclude absorption of BMN 673 (e.g. uncontrolled nausea, vomiting, or diarrhea; malabsorption syndrome; ulcerative disease)
* Absolute neutrophil count >= 1,500/mcL (measured within 28 days prior to entry/ randomization)
* Hemoglobin >= 9 gm/dL (measured within 28 days prior to entry/ randomization)
* Platelets >= 100,000/mcL (measured within 28 days prior to entry/ randomization)
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (measured within 28 days prior to entry/ randomization)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal unless the liver is involved with tumor, in that case, ALT/AST must be =< 5 x upper limit of normal (measured within 28 days prior to entry/ randomization)
* Creatinine clearance >= 50 mL/min (assessed by Cockcroft Gault estimation) (measured within 28 days prior to entry/ randomization)
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Women of child-bearing potential and their partners must agree to use contraception (hormonal or barrier method of birth control; abstinence) from the time of study entry until 30 days after the last dose of study medication; women of child-bearing potential (intact uterus) should have a negative serum pregnancy test; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; female patients must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 consecutive months following cessation of all exogenous hormonal treatments
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation; male partners should be instructed to use contraception during the study period
* Women must not breast-feed while taking the study medications
* Patients must be able to understand and willing to sign an informed consent

Exclusion Criteria:

* Prior treatment for ovarian, fallopian tube, or primary peritoneal cancer
* Receipt of any other investigational agents or any additional anti-cancer agents
* Significant symptom burden from presumed diagnosis including large volume ascites, pain requiring narcotic medication, or shortness of breath on exertion
* Myocardial infarction within 6 months before starting therapy, symptomatic congestive heart failure (New York Heart Association > class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases (e.g., severe hepatic impairment, interstitial lung disease [bilateral, diffuse, parenchymal lung disease], uncontrolled chronic renal diseases [glomerulonephritis, nephritic syndrome, Fanconi syndrome or renal tubular acidosis]), or current unstable or uncompensated respiratory or cardiac conditions, or uncontrolled hypertension (blood pressure >= 140/90), active bleeding diatheses or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus; screening for chronic conditions is not required
* As judged by the investigator, the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Change in deoxyribonucleic acid (DNA) copy number | Baseline to the day of tumor reductive surgery
  Will use descriptive statistics and graphical methods to summarize the change in DNA copy number. Will summarize these changes for untreated patients. Will use a paired t-test to test that mean changes are different from 0. Will test median changes with a Wilcoxon signed-rank test. Will use a 2-sample t-test to compare mean changes between treated and untreated patients. Will compare median changes between treated and untreated patients with a Wilcoxon rank sum test.
Change in ribonucleic acid (RNA) protein expression | Baseline to the day of tumor reductive surgery
  Will use descriptive statistics and graphical methods to summarize the change in RNA protein expression. Will summarize these changes for untreated patients. Will use a paired t-test to test that mean changes are different from 0. Will test median changes with a Wilcoxon signed-rank test. Will use a 2-sample t-test to compare mean changes between treated and untreated patients. Will compare median changes between treated and untreated patients with a Wilcoxon rank sum test. Will use McNemar's test to compare the changes based on homologous recombination deficiency (HRD) assay results.

SECONDARY OUTCOMES:
Overall survival | Up to 3 years
  Will use Cox proportional hazards regression methods to model overall survival as a function of DNA copy number, changes in RNA protein expression, and HRD assay result.
Tumor response | Up to 30 days
  Will use logistic regression methods to model tumor response as a function of changes in DNA copy number, changes in RNA protein expression, and HRD assay result.
Tumor volume | Up to 30 days
  Will use linear regression methods to model tumor volume as a function of changes in DNA copy number, changes in RNA protein expression, and HRD assay result.
Apoptosis | Up to 30 days
  Will use linear regression methods to model apoptosis as a function of changes in DNA copy number, changes in RNA protein expression, and HRD assay result.
Completion Rate of BMN 673 to determine feasibility | Up to 30 days
  Treatment with BMN 673 considered feasible if 70% of patients complete all planned doses of talazoparib and post-operative chemotherapy.
Incidence of adverse events | Up to 30 days
  Will tabulate toxicities by grade and relationship to treatment.
Proportion of patients that exhibit an increase (or decrease) in RNA protein expression greater than 50% | Baseline to the day of tumor reductive surgery
  Will use Fisher's exact test to compare treated and untreated patients with respect to the proportion of patients that exhibit an increase (or decrease) in RNA protein expression. Will compare the mean change in RNA protein expression between those patients with and without a HRD on assay at baseline using a 2-sample t-test. Will compare the median changes between these 2 groups of patients with a Wilcoxon rank sum test. Will compare these 2 groups of patients with respect to HRD assay result using Fisher's exact test.
Change in DNA copy number | Baseline to the day of tumor reductive surgery
  Will use Fisher's exact test to compare treated and untreated patients with respect to the increase (or decrease) in DNA copy number. Will compare the mean change in DNA copy number between those patients with and without a HRD on assay at baseline using a 2-sample t-test. Will compare the median changes between these 2 groups of patients with a Wilcoxon rank sum test. Will compare these 2 groups of patients with respect to HRD assay result using Fisher's exact test.
Change in RNA protein expression | Baseline to the day of tumor reductive surgery
  Will use Fisher's exact test to compare treated and untreated patients with respect to the increase (or decrease) in RNA protein expression. Will compare the mean change in RNA protein expression between those patients with and without a HRD on assay at baseline using a 2-sample t-test. Will compare the median changes between these 2 groups of patients with a Wilcoxon rank sum test. Will compare these 2 groups of patients with respect to HRD assay result using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - M D Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas

REFERENCES:
- [Derived] Sun C, Fang Y, Labrie M, Li X, Mills GB. Systems approach to rational combination therapy: PARP inhibitors. Biochem Soc Trans. 2020 Jun 30;48(3):1101-1108. doi: 10.1042/BST20191092. PMID 32379297
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org